CLINICAL TRIAL: NCT01814774
Title: A Retrospective Chart Review of BOTOX® and Xeomin® for the Treatment of Cervical Dystonia and Blepharospasm
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: TRU2011
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-06

CONDITIONS: Cervical Dystonia; Blepharospasm
MeSH Terms: conditions — Torticollis; Blepharospasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BOTOX®: Retrospective chart review of doses of BOTOX® (onabotulinumtoxinA) used as standard of care in clinical practice. No treatment (intervention) was administered.
  Interventions: Other: No Intervention
- Xeomin®: Retrospective chart review of doses of Xeomin® (incobotulinumtoxinA) used as standard of care in clinical practice. No treatment (intervention) was administered.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No treatment (intervention) was administered.

SUMMARY:
This study is a retrospective chart review to evaluate the doses of botulinum Type A toxins BOTOX® (onabotulinumtoxinA) and Xeomin® (incobotulinumtoxinA) used for the treatment of Cervical Dystonia and Blepharospasm in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* confirmed primary diagnosis of idiopathic cervical dystonia or blepharospasm for at least 2 years
* treatment with Xeomin® and BOTOX® for at least 1 year each

Exclusion Criteria:

* having a neuromuscular junction transmission disorder or taking any medications that could affect neuromuscular junction transmission
* previous surgical procedure involving bone or muscle for the management of cervical dystonia or blepharospasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with cervical dystonia or blepharospasm previously treated with Xeomin® and BOTOX®.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Bergen, Norway
- Wakefield, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Retrospective chart review of doses of BOTOX® (onabotulinumtoxinA) and Xeomin® (incobotulinumtoxinA) used as standard of care in clinical practice. No treatment (intervention) was administered.
Period: Overall Study
Arm/Group | All Participants
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Dose of Botulinum Toxin Used to Treat Cervical Dystonia
Description: The average dose of botulinum toxin received per patient per year was calculated.
Time Frame: 2 Years
Population: Participants diagnosed with Cervical Dystonia who received onabotulinumtoxinA for 2 years and incobotulinumtoxinA for 2 years.
Measure: Mean (95% Confidence Interval); unit: units per patient per year
Arm/Group | BOTOX® | Xeomin®
Number analyzed (Participants) | 25 | 25
units per patient per year | 444.70 [347.16 to 542.24] | 536.30 [409.64 to 662.96]

2. Primary Outcome: Dose of Botulinum Toxin Used to Treat Blepharospasm
Description: The average dose of botulinum toxin received per patient per year was calculated.
Time Frame: 2 Years
Population: Participants diagnosed with Blepharospasm who received onabotulinumtoxinA for 2 years and incobotulinumtoxinA for 2 years.
Measure: Mean (95% Confidence Interval); unit: units per patient per year
Arm/Group | BOTOX® | Xeomin®
Number analyzed (Participants) | 14 | 14
units per patient per year | 50.40 [21.21 to 79.59] | 64.01 [33.32 to 94.70]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: An Adverse Event was any unfavorable and unintended sign, symptom, or disease documented in the medical chart that occurred after treatment with botulinum toxin, or pre-existing conditions that worsened during the retrospective period.
Time Frame: 2 Years
Population: Safety population included all participants who received at least one dose of botulinum toxin.
Measure: Number; unit: participants
Arm/Group | BOTOX® | Xeomin®
Number analyzed (Participants) | 48 | 48
participants | 12 | 10

4. Secondary Outcome: Botulinum Toxin Inter-injection Interval
Description: Injection-interval was the time in weeks between injections of botulinum toxin.
Time Frame: 2 Years
Population: All participants who received onabotulinumtoxinA for 2 years and incobotulinumtoxinA for 2 years.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | BOTOX® | Xeomin®
Number analyzed (Participants) | 39 | 39
weeks | 15.83 (4.02) | 14.39 (3.38)

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | BOTOX® | Xeomin®
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 7/48 | 4/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® (N=48) | Xeomin® (N=48)
Dysphagia (Gastrointestinal disorders) | 4 | 1
Ptosis (Eye disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.